CLINICAL TRIAL: NCT00907517
Title: A Phase 1 Dose-Escalation Study of SCH 900776 in Combination With Cytarabine in Subjects With Acute Leukemias (Protocol No. P05247)
Brief Title: Study of SCH 900776 (MK-8776) With and Without Cytarabine in Participants With Acute Leukemias (P05247)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P05247; MK-8776-001 (Other: Merck Protocol Number)
Record Dates: First submitted 2009-05-21; First posted 2009-05-22 (Estimated); Results first posted 2017-01-25 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Myelogenous Leukemia, Acute; Leukemia, Lymphocytic, Acute; Leukemia, Lymphoblastic, Acute, Philadelphia-Positive; Myelogenous Leukemia, Chronic, Aggressive Phase
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Accelerated Phase | interventions — MK-8776; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- MK-8776 10 mg/m^2 + Cytarabine 2 g/m^2 (Experimental): Participants received MK-8776 10 mg/m^2 intravenously (IV) on Days 2 and 3 and again on Days 11 and 12 PLUS cytarabine 2 g/m^2 IV via 72-hour continuous intravenous infusion (CIV) on Days 1 through 3 and repeated on Days 10 through 12 of a treatment cycle. The duration of one treatment cycle was to be approximately 4 to 6 weeks (until hospital discharge).
  Interventions: Drug: MK-8776; Drug: Cytarabine
- MK-8776 20 mg/m^2 + Cytarabine 2 g/m^2 (Experimental): Participants received MK-8776 20 mg/m^2 IV on Days 2 and 3 and again on Days 11 and 12 PLUS cytarabine 2 g/m^2 IV via 72-hour CIV on Days 1 through 3 and repeated on Days 10 through 12 of a treatment cycle. The duration of one treatment cycle was to be approximately 4 to 6 weeks (until hospital discharge).
  Interventions: Drug: MK-8776; Drug: Cytarabine
- MK-8776 40 mg/m^2 + Cytarabine 2 g/m^2 (Experimental): Participants received MK-8776 40 mg/m^2 IV on Days 2 and 3 and again on Days 11 and 12 PLUS cytarabine 2 g/m^2 IV via 72-hour CIV on Days 1 through 3 and repeated on Days 10 through 12 of a treatment cycle. The duration of one treatment cycle was to be approximately 4 to 6 weeks (until hospital discharge).
  Interventions: Drug: MK-8776; Drug: Cytarabine
- MK-8776 56 mg/m^2 + Cytarabine 2 g/m^2 (Experimental): Participants received MK-8776 56 mg/m^2 IV on Days 2 and 3 and again on Days 11 and 12 PLUS cytarabine 2 g/m^2 IV via 72-hour CIV on Days 1 through 3 and repeated on Days 10 through 12 of a treatment cycle. The duration of one treatment cycle was to be approximately 4 to 6 weeks (until hospital discharge).
  Interventions: Drug: MK-8776; Drug: Cytarabine
- MK-8776 140 mg + Cytarabine 2 g/m^2 (Experimental): Participants received MK-8776 140 mg flat dose IV on Days 2 and 3 and again on Days 11 and 12 PLUS cytarabine 2 g/m^2 IV via 72-hour CIV on Days 1 through 3 and repeated on Days 10 through 12 of a treatment cycle. The duration of one treatment cycle was to be approximately 4 to 6 weeks (until hospital discharge).
  Interventions: Drug: MK-8776; Drug: Cytarabine

INTERVENTIONS:
Drug: MK-8776 — IV infusion
  Other Names: SCH 900776
Drug: Cytarabine — IV infusion
  Other Names: Generic: ara-C and cytosine arabinoside; Cytosar-U®

SUMMARY:
This study of SCH 900776 (MK-8776) will evaluate its safety and tolerability when given in combination with cytarabine to participants with acute leukemias. Participants in the Dose-Escalation Part will be enrolled in cohorts that will receive sequentially higher doses of MK-8776 in combination with standard doses of cytarabine. Only one combination treatment cycle of approximately 4 to 6 weeks is anticipated, but participants may receive additional cycles if clinically indicated after discussion between the Investigator and the Sponsor. The recommended combination doses for a Phase 2 trial (RP2D) will be determined based on safety and biological activity. Up to 10 to 15 additional participants will be studied at the combination RP2D.

ELIGIBILITY:
Inclusion Criteria:

* Must have a histologically or cytologically confirmed diagnosis of relapsed and/or refractory acute leukemia, including:

  * acute myelogenous leukemia (AML), including AML arising from myelodysplasia (MDS) or myeloproliferative disorder (MPD);
  * acute lymphocytic leukemia, including Philadelphia chromosome-positive (Ph+) ALL (Dose-Escalation Part only);
  * chronic myelogenous leukemia (CML) in accelerated phase (AP) or blast crisis (BC) of either myeloid or lymphoid origin (Dose-Escalation Part only);
  * treatment-related high-grade MDS (i.e. refractory anemia with excess blasts in transformation [RAEBT]);
  * MPD in transformation [eg, CMMoL-T (5%-19% blasts)].
* Must have recurred or progressed following standard therapy or failed standard therapy, or have disease for which no standard therapy currently exists.
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Females of childbearing potential must have a negative pregnancy test within 5 days prior to first dose of cytarabine.
* Females of childbearing potential and males whose sexual partner is of childbearing potential must agree to abstain from sexual intercourse or to use an acceptable method of contraception during the study and for 90 days following the last dose of study treatment.
* Must have adequate renal function as evidenced by a serum creatinine level <=1.5 x upper limit of normal (ULN) or a calculated creatinine clearance >=60 mL/min.
* Participants, except ones with known Gilbert's Syndrome, must have adequate hepatic function as evidenced by a serum bilirubin level <=1.5 mg/dL AND serum levels of aspartate and alanine aminotransferase (AST/ALT) <=5 x the ULN for the reference laboratory.
* Must have adequate cardiac function with a left ventricular ejection fraction (LVEF) of >=45% (echocardiogram or multiple-gated acquisition [MUGA] scan).
* Must be recovered from the effects of any prior surgery, radiotherapy, or systemic antineoplastic therapy.
* Participants who are refractory to or relapsed after prior allogeneic or autologous stem cell transplant are eligible.

Exclusion Criteria:

* Must not have known hypersensitivity to MK-8776 or cytarabine or to any of their excipients or have received therapy with another Checkpoint kinase 1 (CHK1) inhibitor.
* Must not have persistent, unresolved Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v 3.0) ≥ Grade 2 drug-related toxicity (except alopecia, erectile impotence, hot flashes, decreased libido, hematologic toxicity) associated with previous treatment.
* Must not have known human immunodeficiency virus (HIV), hepatitis B or hepatitis C, or have a known history of liver cirrhosis or active alcohol abuse.
* Must not be New York Heart Association (NYHA) Class III (has marked limitation in activity due to symptoms, even during less than ordinary activity [e.g. walking short distances >20-100 m]; is comfortable only at rest) or Class IV (has severe limitations; experiences symptoms even while at rest; mostly bed bound).
* Must not have undergone major surgery within 3 weeks prior to first study drug administration after enrollment.
* Must not have known active central nervous system (CNS) or leptomeningeal leukemia.
* Must not have received radiation therapy within 2 weeks prior to first study treatment administration after enrollment or radiation therapy to >25% of bone marrow.
* Must not have received more than 4 prior induction regimens.
* Must not have a peripheral blast count ≥50,000/mm^3.
* Must not have active, uncontrolled graft versus host disease (GVHD) post-allogeneic stem cell transplant.
* Must not have had any of the following within 6 months prior to first study treatment administration after enrollment: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or seizure disorder.
* Must not have a known bleeding diathesis, e.g. hemophilia, or disseminated intravascular coagulation.
* Must not have an active, uncontrolled infection.
* Must not have a history of cytarabine-related neurotoxicity.
* Must not have a baseline corrected QT (QTc) interval >470 msec (i.e. CTCAE v 3.0 Grade ≥2).
* Must not currently be a smoker and/or must not be likely to smoke during the study.
* Females must not be breast-feeding, pregnant, or intend to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-07-29 (Actual); Primary Completion 2011-06-13 (Actual); Study Completion 2011-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Karp JE, Thomas BM, Greer JM, Sorge C, Gore SD, Pratz KW, Smith BD, Flatten KS, Peterson K, Schneider P, Mackey K, Freshwater T, Levis MJ, McDevitt MA, Carraway HE, Gladstone DE, Showel MM, Loechner S, Parry DA, Horowitz JA, Isaacs R, Kaufmann SH. Phase I and pharmacologic trial of cytosine arabinoside with the selective checkpoint 1 inhibitor Sch 900776 in refractory acute leukemias. Clin Cancer Res. 2012 Dec 15;18(24):6723-31. doi: 10.1158/1078-0432.CCR-12-2442. Epub 2012 Oct 23. PMID 23092873

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only one combination treatment cycle of approximately 4 to 6 weeks duration was anticipated, but participants may have received additional cycles of treatment if clinically indicated after discussion between the Investigator and the Sponsor.
Period: Overall Study
Arm/Group | MK-8776 10 mg/m^2 + Cytarabine 2 g/m^2 | MK-8776 20 mg/m^2 + Cytarabine 2 g/m^2 | MK-8776 40 mg/m^2 + Cytarabine 2 g/m^2 | MK-8776 56 mg/m^2 + Cytarabine 2 g/m^2 | MK-8776 140 mg + Cytarabine 2 g/m^2
Started | 3 | 3 | 6 | 6 | 6
Completed | 0 | 0 | 2 | 2 | 1
Not Completed | 3 | 3 | 4 | 4 | 5
Not completed — Progressive Disease | 3 | 3 | 4 | 4 | 4
Not completed — Symptomatic Deterioration | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- MK-8776 10 mg/m^2 + Cytarabine 2 g/m^2: Participants received MK-8776 10 mg/m^2 IV on Days 2 and 3 and again on Days 11 and 12 PLUS cytarabine 2 g/m^2 IV via 72-hour CIV on Days 1 through 3 and repeated on Days 10 through 12 of a treatment cycle. The duration of one treatment cycle was to be approximately 4 to 6 weeks (until hospital discharge).
- Total: Total of all reporting groups
Arm/Group | MK-8776 10 mg/m^2 + Cytarabine 2 g/m^2 | MK-8776 20 mg/m^2 + Cytarabine 2 g/m^2 | MK-8776 40 mg/m^2 + Cytarabine 2 g/m^2 | MK-8776 56 mg/m^2 + Cytarabine 2 g/m^2 | MK-8776 140 mg + Cytarabine 2 g/m^2 | Total
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.3 (9.1) | 55.7 (1.5) | 44.2 (14.2) | 57.5 (18.3) | 56.3 (13.5) | 53.9 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 2 | 4 | 3 | 13
  Male | 2 | 0 | 4 | 2 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Dose-limiting Toxicity (DLT)
Description: Toxicity was assessed according to the Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v 3.0). DLTs in Cycle 1 consisted of any of the following: 1) Selected Grade 4 drug-related nonhematologic toxicities, 2) Selected Grade 3 drug-related nonhematologic toxicities that do not resolve to ≤ Grade 2 within 48 hours: Neurotoxicity of any duration, Nephrotoxicity of any duration, QT interval corrected by Fridericia (QTcF) prolongation of any duration, 3) Inability to administer Day 10 cytarabine therapy due to ongoing, uncontrolled serious or life-threatening toxicity. The number of participants who experienced a DLT during Cycle 1 is summarized.
Time Frame: Throughout Cycle 1 (Up to 6 weeks)
Population: The population consisted of all participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | MK-8776 10 mg/m^2 + Cytarabine 2 g/m^2 | MK-8776 20 mg/m^2 + Cytarabine 2 g/m^2 | MK-8776 40 mg/m^2 + Cytarabine 2 g/m^2 | MK-8776 56 mg/m^2 + Cytarabine 2 g/m^2 | MK-8776 140 mg + Cytarabine 2 g/m^2
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 3

2. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. An AE can be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a study treatment, whether or not considered related to this study treatment. The number of participants who experienced an AE is summarized.
Time Frame: Up to 45 days after last dose of study treatment (Up to 180 days)
Population: The population consisted of all participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | MK-8776 10 mg/m^2 + Cytarabine 2 g/m^2 | MK-8776 20 mg/m^2 + Cytarabine 2 g/m^2 | MK-8776 40 mg/m^2 + Cytarabine 2 g/m^2 | MK-8776 56 mg/m^2 + Cytarabine 2 g/m^2 | MK-8776 140 mg + Cytarabine 2 g/m^2
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 6
Participants | 3 | 3 | 6 | 6 | 6

3. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. An AE can be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a study treatment, whether or not considered related to this study treatment. The number of participants who discontinued study treatment due to an AE is summarized.
Time Frame: Up to 135 days
Population: The population consisted of all participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | MK-8776 10 mg/m^2 + Cytarabine 2 g/m^2 | MK-8776 20 mg/m^2 + Cytarabine 2 g/m^2 | MK-8776 40 mg/m^2 + Cytarabine 2 g/m^2 | MK-8776 56 mg/m^2 + Cytarabine 2 g/m^2 | MK-8776 140 mg + Cytarabine 2 g/m^2
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 45 days after last dose of study treatment (Up to 180 days)
Description: The population consisted of all participants who received at least one dose of study treatment.
Arm/Group | MK-8776 10 mg/m^2 + Cytarabine 2 g/m^2 | MK-8776 20 mg/m^2 + Cytarabine 2 g/m^2 | MK-8776 40 mg/m^2 + Cytarabine 2 g/m^2 | MK-8776 56 mg/m^2 + Cytarabine 2 g/m^2 | MK-8776 140 mg + Cytarabine 2 g/m^2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 1/6 | 2/6 | 1/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8776 10 mg/m^2 + Cytarabine 2 g/m^2 (N=3) | MK-8776 20 mg/m^2 + Cytarabine 2 g/m^2 (N=3) | MK-8776 40 mg/m^2 + Cytarabine 2 g/m^2 (N=6) | MK-8776 56 mg/m^2 + Cytarabine 2 g/m^2 (N=6) | MK-8776 140 mg + Cytarabine 2 g/m^2 (N=6)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FUNGAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA FUNGAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8776 10 mg/m^2 + Cytarabine 2 g/m^2 (N=3) | MK-8776 20 mg/m^2 + Cytarabine 2 g/m^2 (N=3) | MK-8776 40 mg/m^2 + Cytarabine 2 g/m^2 (N=6) | MK-8776 56 mg/m^2 + Cytarabine 2 g/m^2 (N=6) | MK-8776 140 mg + Cytarabine 2 g/m^2 (N=6)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0)
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 5 (6) | 3 (5) | 5 (7)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (4) | 1 (1) | 1 (1) | 2 (4) | 0 (0)
SPLENOMEGALY (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (16) | 1 (1) | 1 (6) | 1 (3) | 1 (2)
CARDIOMEGALY (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
EXTRASYSTOLES (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
TRICUSPID VALVE INCOMPETENCE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EAR PAIN (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOACUSIS (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIABETES INSIPIDUS (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
CONJUNCTIVITIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DRY EYE (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PERIORBITAL OEDEMA (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VISUAL IMPAIRMENT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL TENDERNESS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4) | 4 (6) | 2 (3)
DRY MOUTH (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EPIGASTRIC DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
MELAENA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (2) | 1 (1) | 4 (7) | 5 (5) | 5 (6)
OESOPHAGEAL ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PROCTALGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SALIVARY HYPERSECRETION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (7) | 4 (4) | 1 (1)
CATHETER SITE ERYTHEMA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHILLS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 3 (3)
MALAISE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
MUCOSAL INFLAMMATION (General disorders) | 2 (12) | 1 (1) | 2 (3) | 4 (5) | 0 (0)
NODULE (General disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
OEDEMA (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 1 (2)
PAIN (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 2 (9) | 2 (2) | 0 (0)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 2 (8) | 1 (1) | 2 (12) | 1 (3) | 2 (2)
BACTERAEMIA (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
CANDIDIASIS (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
CELLULITIS ORBITAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
FUNGAEMIA (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
MASTOIDITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
PNEUMONIA FUNGAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TINEA INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TOOTH ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
EYE INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PERIORBITAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 1 (1) | 3 (10) | 2 (7) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1) | 3 (8) | 2 (9) | 0 (0)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 (3) | 1 (3) | 2 (6) | 4 (5) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLOOD CREATININE DECREASED (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 0 (0) | 2 (2) | 3 (5) | 1 (3)
CARDIAC MURMUR (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EJECTION FRACTION DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
FUNGAL TEST POSITIVE (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
TROPONIN INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
WEIGHT DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FLUID OVERLOAD (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
FLUID RETENTION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (6) | 0 (0)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (4) | 2 (7) | 1 (3)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (4)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
HYPOPHAGIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 1 (1) | 3 (5) | 2 (3) | 1 (1)
MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABNORMAL DREAMS (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AGITATION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
DELIRIUM (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HALLUCINATION, AUDITORY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INSOMNIA (Psychiatric disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (2)
BLADDER PAIN (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CYSTITIS HAEMORRHAGIC (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DYSURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INCONTINENCE (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEPHROGENIC DIABETES INSIPIDUS (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEUROGENIC BLADDER (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BREAST CYST (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
NASAL DRYNESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
PARANASAL SINUS HYPERSECRETION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (2)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN MASS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (10) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the study.